CLINICAL TRIAL: NCT04288596
Title: The Canadian Registry for Adults With Congenital Heart Disease Interventions
Brief Title: Canadian Adult Congenital Heart Disease Intervention Registry
Acronym: C-ACHDiR
Status: Not yet recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Eric Horlick, Interventional and Congenital Cardiologist, University Health Network, Toronto
Other Study IDs: CRegistry
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Atrial Septal Defect; Patent Foramen Ovale; Tetralogy of Fallot; Fontan; Coarctation of Aorta; Transposition of Great Vessels; Percutaneous Pulmonary Valve Implantation
MeSH Terms: conditions — Heart Septal Defects, Atrial; Foramen Ovale, Patent; Tetralogy of Fallot; Aortic Coarctation; Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eligible for Registry: All consecutive patients who undergo any of the five ACHDi interventions (complex catheterization, ASD closure, PFO closure, CoA stenting, and PPVI) at the time of Registry launch, who have also consented to participate.
  Interventions: Other: Participants undergoing ACHD intervention

INTERVENTIONS:
Other: Participants undergoing ACHD intervention — Participants will receive standard of care for their ACHD intervention.

SUMMARY:
The ACHDi Registry study will create a foundational database for adult congenital heart disease interventions. This Pan-Canadian Registry will collect clinical and patient-reported information that will enable the evaluation of care processes and outcomes in five most common ACHDi interventions by enabling prospective and retrospective registry-based studies to answer important clinical practice and policy-relevant questions.

DETAILED DESCRIPTION:
The goal of this study is to establish a rigorously developed registry to enable an impactful research agenda in adults with congenital heart disease interventions (ACHDi). The clinical and patient-reported information captured in the Registry will allow researchers to evaluate care processes and outcomes in five most common ACHDi interventions including transcatheter closure of atrial septal defects, closure of patent foramen ovale, coarctation of aorta stenting, percutaneous pulmonary valve implantation, and complex catheterization.

In 2019, we established the Canadian Research Network for ACHD Interventions (CRN-ACHDi), a national ACHD research network bringing together researchers, providers, patients, and policymakers from 4 provinces (Alberta, British Columbia, Ontario and Quebec) to improve patient experiences and outcomes through i) a national registry with modern data platform; ii) a rigorously established national research priorities agenda; and iii) a strong collaborative and multidisciplinary research environment.

The C-ACHDi Registry will provide opportunities for researchers to ask clinical practice and policy-relevant research questions that are supported by high quality data. In addition, it will provide an opportunity for patients to contribute data for meaningful and high quality clinical and translational research. The C-ACHDi Registry will provide a base for conducting registry-based studies (e.g., prospective experimental, prospective and retrospective observational) in the future as well as a foundation for benchmark and quality improvement activities.

ELIGIBILITY:
Inclusion Criteria:

* participants must be 18 years or older referred for intervention for one of five ACHD conditions including diagnostic catheterization for complex ACHD patients (Tetralogy of Fallot, Fontan, and transposition of the great vessels, single ventricle, truncus arteriosus); transcatheter closure of atrial septal defects; transcatheter closure of patent foramen ovale; coarctation of aorta stenting, and percutaneous pulmonary valve implantation.

Exclusion Criteria:

* participants below the age of 18
* participants residing outside of Canada

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes all consecutive patients who undergo any of the five ACHDi interventions (complex catheterization, ASD closure, PFO closure, CoA stenting, and PPVI) from the time of launching the registry (April 1, 2020 as the tentative starting date), and consent to participate in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
the number of subjects enrolled | baseline
  This is an observational registry. The primary outcome is the number of subjects enrolled who are undergoing ACHD intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Horlick, MD, Principal Investigator — University Health Network, Peter Munk Cardiac Centre; Lusine Abrahamyan, MD, PhD, Principal Investigator — University Health Network, Theta Collaborative
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient health card numbers will be collected to be linked with Canadian Healthcare administrative databases.